CLINICAL TRIAL: NCT00357305
Title: Phase I Study of Vorinostat (Suberoylanilide Hydroxamic Acid, or SAHA) in Combination With Cytosine Arabinoside (Ara-C) and Etoposide for Patients With Relapsed and/or Refractory Acute Leukemias, Myelodysplasias and Myeloproliferative Disorders
Brief Title: Vorinostat, Cytarabine, and Etoposide in Treating Patients With Relapsed and/or Refractory Acute Leukemia or Myelodysplastic Syndromes or Myeloproliferative Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00088; GCC 0447; NCI-6829; CDR0000487484
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Acute Promyelocytic Leukemia (M3); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; de Novo Myelodysplastic Syndromes; Essential Thrombocythemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Polycythemia Vera; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Myeloproliferative Disorders; Polycythemia Vera; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vorinostat; Cytarabine; Etoposide

ARMS (1):
- Treatment (enzyme inhibitor, chemotherapy) (Experimental): Patients receive oral SAHA two or three times daily on days 1-7 and cytarabine IV over 3 hours twice daily and etoposide IV over 1 hour once daily on days 11-14. Treatment repeats approximately every 6-7 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: cytarabine; Drug: etoposide; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with cytarabine and etoposide in treating patients with relapsed or refractory acute leukemia or myelodysplastic syndromes or myeloproliferative disorders. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving vorinostat together with cytarabine and etoposide may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the feasibility, tolerability, and toxicities, in terms of the maximum tolerated dose (MTD), of the sequential combination of vorinostat (SAHA) followed by cytarabine and etoposide in patients with relapsed and/or refractory acute leukemia or transforming myelodysplastic syndromes or myeloproliferative disorders.

II. Determine whether the addition of SAHA to cytarabine and etoposide chemotherapy improves outcome, in terms of complete response rate, duration of response, and overall survival, in these patients.

III. Determine the effects of SAHA on induction of tumor necrosis factor-related apoptosis-inducing ligand (TRAIL)-death receptors DR4 and DR5 and other pro-apoptotic mediators in patient-derived cancer cells (leukemia blast cells) and somatic cells (buccal mucosa cells, using pre-SAHA and on SAHA treatment samples).

IV. Determine the ability of SAHA to block leukemia blast cells in the G1 phase of the cell cycle (leukemia blast cells, using pre-SAHA and on SAHA treatment samples).

V. Determine the effects of SAHA on the expression of P-glycoprotein/MDR1/ABCB1, and the breast cancer resistance protein (BCRP/ABCG2), using functional and mRNA/protein assays for these transporters (leukemia blast cells, using pre-SAHA and on SAHA treatment samples).

OUTLINE: This is a dose-escalation study of vorinostat (SAHA).

Patients receive oral SAHA two or three times daily on days 1-7 and cytarabine intravenously (IV) over 3 hours twice daily and etoposide IV over 1 hour once daily on days 11-14. Treatment repeats approximately every 6-7 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients who achieve complete response after 1 course of therapy may receive 1 or 2 more courses of therapy. Patients who achieve partial response after 1 course of therapy may receive 1 more course of therapy. Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 10 patients are treated at that dose. Blood, buccal cells, and bone marrow samples are collected prior to and during treatment. Samples are used for pharmacokinetic and pharmacodynamic studies, protein expression studies, and gene expression profiling. After completion of study treatment, patients are followed within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Relapsed or refractory acute myeloid leukemia (AML)

    * Patients with acute promyelocytic leukemia t(15;17) must have failed prior tretinoin and arsenic trioxide-containing regimen

      * Must be refractory to both agents with absence of durable hematologic response OR relapsed after a complete response duration of < 6 months
  * Relapsed or refractory acute lymphoblastic leukemia
  * Chronic myelogenous leukemia in accelerated or blastic phase

    * Must be refractory to treatment with imatinib mesylate or dasatinib

      * Disease progression despite continued treatment with imatinib mesylate or dasatinib
    * Patients in accelerated or blastic phase are eligible if unable to tolerate imatinib mesylate provided their disease has progressed on dasatinib or if unable to tolerate dasatinib
  * AML arising in the setting of underlying myelodysplastic syndromes (MDS) and/or myeloproliferative disorders (MPD)
  * Secondary or therapy-related AML
* No active CNS leukemia
* Leukostasis OR leukemic blast count > 50,000/mm³ allowed provided patient is treated with emergency leukapheresis or hydroxyurea to reduce leukemic blast count to < 30,000/mm³
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of cytarabine-related neurotoxicity
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat (SAHA) or other agents used in the study
* No other uncontrolled illness, including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude compliance with study requirements
* Infection allowed provided patient is receiving active treatment
* No HIV positivity
* See Disease Characteristics
* Recovered from prior therapy

  * Persistent alopecia, fingernail discoloration, or hematologic abnormalities (primarily related to underlying disease) > 4 weeks after last course of chemotherapy or radiotherapy does not exclude patient
* At least 2 weeks since prior valproic acid or any other histone deacetylase inhibitor
* No more than 3 prior courses of induction/reinduction chemotherapy, including induction and consolidation therapy or induction therapy after any bone marrow transplantation or similar procedure

  * Prior low-dose azacitidine, growth factors, cytokines, thalidomide, interferon, or imatinib mesylate for treatment of preceding MDS/MPD do not count as prior induction/reinduction therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas [e.g., carmustine] or mitomycin C) or radiotherapy
* At least 24 hours since prior hydroxyurea
* At least 2 weeks since prior imatinib mesylate, hematopoietic growth factors, and biological agents
* At least 4 weeks since prior autologous stem cell transplantation
* Prior allogeneic stem cell transplantation allowed if all of the following criteria are met:

  * At least 90 days since prior transplant
  * No evidence of graft-vs-host disease
  * At least 2 weeks since prior immunosuppressive therapy
* No other concurrent anticancer agents or therapies
* No other concurrent investigational agents
* Concurrent hydroxyurea or leukapheresis allowed on days 1-10 of study treatment to control rising leukemic blasts (blasts > 30,000/mm³) or leukostasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-05; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of vorinostat (SAHA) in combination with cytarabine and etoposide | Course 1
  Based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Response rate | Baseline, day 4-7 of course 1, and after each course
  Measured using a bone marrow aspirate and/or biopsy. 90% confidence interval will be calculated
Progression-free survival | At 30 days after completion of study treatment and continued follow up visits
  Estimated using the Kaplan-Meir method.
Disease-specific survival | At 30 days after completion of study treatment and continued follow up visits
  Estimated using the Kaplan-Meir method.
One-year survival | At 1 year
  Estimated using the Kaplan-Meir method.
Overall survival | At 30 days after completion of study treatment and continued follow up visits
  Measured from time of enrollment onto this study to the time of death. Estimated using the Kaplan-Meir method.
Degree of upregulation of tumor necrosis factor-related apoptosis-inducing ligand (TRAIL)-death receptors and proteins associated with apoptosis | Baseline and days 4-7 of course 1
  Performed by the Rnase protection assay.
Alterations in cell cycle phase | Baseline and days 4-7 of course 1
  Patient-derived bone marrow or peripheral blood mononuclear cells will be evaluated for cell cycle phase distribution, using the hypotonic propidium-iodide method and flow cytometry.
Expression of MDR proteins at MTD of SAHA | Baseline and days 4-7 of course 1
  Using quantitative, real-time polymerase chain reaction (PCR) methods with product detected using specific hybridization probes.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Ross, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (2):
- United States (2):
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania